CLINICAL TRIAL: NCT03443505
Title: Pilot Feasibility Study to Determine the Clinical Effectiveness of Neural Respiratory Drive (NRD) to Predict COPD Exacerbations at Home.
Brief Title: NRD to Predict COPD Exacerbations at Home
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 232384
Record Dates: First submitted 2018-02-09; First posted 2018-02-23 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; Acute exacerbation; Neural respiratory drive; Parasternal electromyography; Respiratory physiology; Lung function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Neural respiratory drive measurement — Neural respiratory drive (NRD) has been validated as an objective physiological biomarker in acute exacerbation of chronic obstructive pulmonary disease (AECOPD). Change in NRD during hospital admission has been demonstrated to be a marker of physician-defined clinical deterioration. NRD is a non-invasive measurement that involves skin preparation with a gel and alcohol wipe before placing 3 surface electrodes on the chest wall and collar bone to perform electromyography (EMG) of parasternal muscles. Electrodes are connected to an automated EMG analysis system to derive a measurement of NRD. Measurements take approximately 10 minutes with subject being monitored during normal ("tidal") breathing and performing maximal sniff manoeuvres.

SUMMARY:
COPD is a common, serious disease and is a major burden on patients and the National Health Service. Patients with COPD can develop worsening of their symptoms, known as an exacerbation, which can be severe enough to warrant hospital admission. There are currently no objective measurements available to patients and clinicians to predict exacerbation and monitor recovery. Detection of exacerbation by both patients and physicians is known to correlate poorly with onset of respiratory deterioration.

Measurement of neural respiratory drive (NRD), or drive to breathe, using respiratory muscle electromyography (EMG) correlates with changes in patients' symptoms and physician defined deterioration during hospital admissions.

This pilot study aims to identify whether daily measurement of NRD at home following admission to hospital with exacerbation of COPD can detect an exacerbation within 30 days of discharge (20% of patients are readmitted within this period). This technique could enable early detection of deterioration at home, facilitating earlier treatment compared to current practice, potentially avoiding hospital readmission.

30 patients admitted to St Thomas' Hospital because of an exacerbation of COPD aged 40-80, with a body mass index <35kg/m2, who can follow English instructions and give informed consent, who are discharged home will be recruited. If patients consent to participate, they will have assessments as inpatients and for 30 days at home following discharge, or until hospital readmission, whichever is sooner. Assessments include vital observations (heart rate, blood pressure, respiratory rate and oxygen saturations), NRD, and a symptom questionnaire. At the baseline assessment, age, height weight, a brief medical history, results of tests already taken by the clinical team (blood tests and chest x-ray) and lung function tests will be recorded. This study will take 12 months. Philips and its Affiliates are providing the NRD measuring equipment.

DETAILED DESCRIPTION:
Introduction

COPD is a common and serious disease, and is a major burden on patients and the National Health Service. Current markers to detect and monitor exacerbations and response to treatment are based on symptoms reported by patients, clinical assessment and Early Warning Scores, which are a composite measurement of standard observations, including heart rate, blood pressure, respiratory rate and oxygen saturations. However these scores have been validated on general populations and there is concern regarding their application to COPD patients. There is currently no objective biomarker to predict and monitor COPD exacerbations in routine clinical use.

NRD is measured using parasternal intercostal EMG measurements. Daily NRD measurements during hospital admission with exacerbation of COPD has been demonstrated to be a reproducible non-invasive measurement which is acceptable to patients. Importantly, it can reliably detect clinical deterioration and worsening in patient reported breathlessness more reliably than current standard assessments.

This observational pilot feasibility study is designed to identify whether NRD can be measured reliably at home following discharge from hospital with exacerbation of COPD, and whether it can detect respiratory deterioration within 30 days. This technique thus has the potential to allow early detection of deterioration at home, which can facilitate early treatment in the community and potentially avoid hospital readmission, which would have a profound impact on both patients and the NHS.

Study objectives

Primary: The primary objective of the study is to investigate whether home measurement of NRD can detect an exacerbation of COPD (symptom based definition) within a 30-day post hospital discharge period.

Secondary

Clinical:

* To validate NRD as an advanced physiological biomarker of clinical respiratory deterioration and a re-exacerbation of COPD
* To analyse NRD trajectory as it relates to standardly subjective measurements of respiratory symptoms e.g. COPD Assessment Test (CAT) and Modified Borg Scale (mBorg), or symptoms as assessed by the EXACT-PRO questionnaire
* To determine positive and negative predictive value of NRD, and/or a combination of clinical features, to detect clinical respiratory deterioration
* To assess correlation of change in NRD, physical activity and symptom resolution

Feasibility:

-To investigate quality of parasternal EMG measurements performed in the home environment

Technical:

-To use the data collected during the study to tune, refine, optimise the automated NRD calculation algorithm

Study end-points Primary end-point: Change in NRD from baseline to day prior to an acute exacerbation of COPD.

Secondary outcomes

* Change in NRD from peak exacerbation (hospital) to recovery baseline (home)
* Correlation of time to recovery as measured by NRD and EXACT-PRO
* Correlation of NRD to EXACT-PRO from hospital discharge to recovery
* Correlation of NRD to physical activity from hospital discharge to recovery
* Physician-assessed exacerbation within 30-day post-discharge
* Self-treated exacerbation within 30-day post-discharge
* All cause hospital readmission within 30-day post-discharge
* Mortality within 30-day post-discharge
* Recovery as defined by the EXACT-PRO within 30-day post-discharge
* Medication change within 30-day post-discharge
* Unplanned healthcare contacts
* Attendance of emergency department (without admission)

Methods

30 consecutive patients admitted to St Thomas' Hospital with a primary diagnosis of exacerbation of COPD will be enrolled within 16 hours of admission who fulfil inclusion and exclusion criteria (listed below). Baseline assessments will include recording of age, height, weight, pack year smoking history, exacerbation frequency, pre-admission lung function and breathlessness score, co-morbidities, regular medications, chest x-ray, venous and arterial blood test results already taken by the medical team, symptom questionnaires (CAT, mBorg and EXACT-PRO), vital observations (heart rate, blood pressure, respiratory rate, oxygen saturation and use of supplementary oxygen), lung function and NRD. Participants will receive inpatient assessments by an investigator to receive an update from the clinical team and measure standard observations, NRD and complete the EXACT-PRO questionnaire. On the day of discharge, participants' updated medical history and blood tests will be documented and vital observations, symptom questionnaires (CAT, mBorg and EXACT-PRO), lung function and NRD will be measured. Participants will be issued with a physical activity monitor which will be worn for the remaining duration of the study. Participants will then receive home visits from an investigator, who are experienced in the management of COPD, to measure NRD, complete the EXACT-PRO symptom questionnaire and review participants' daily symptom diary. Lung function and the CAT symptom questionnaire will be performed weekly at home. Participants will be followed up for 30 days following hospital discharge or until they are readmitted to hospital, whichever is sooner.

Study design: Observational cohort design

Inclusion criteria

* Age 40-80 years
* Patients hospitalised with a primary diagnosis of an acute exacerbation of COPD
* Body mass index (BMI) ≤ 35 kg/m2
* Cognitively and linguistically able to follow instructions given in English and provide informed consent
* To be discharged to home following the hospitalisation
* Patient lives in the catchment area served by the Integrated Respiratory Team at Guy's and St Thomas' NHS Foundation Trust in a home environment deemed safe by the investigators to perform home assessments

Exclusion criteria

* Previous home PAP (CPAP or NIV) therapy use within the past year, or post-discharge
* Allergies to latex, metals or local anaesthetic agents
* Wound or inflamed skin at parasternal location (2nd intercostal space)
* History of skin allergies or sensitivity to cosmetics and lotions
* Psychological and social factors that would impair compliance with study protocol and schedule
* Any major non-COPD chronic disease or condition, such as severe heart failure (LVEF<30%), malignancy (active treatment and palliation), end stage renal failure/dialysis, significant neuromuscular disease (eg. NMD, MD) determined by review of medical history and / or patient reported medical history that may contribute significantly to risk of readmission, as determined by PI
* Length of stay < 6 hours
* Planned travel away from home within the 30 day post discharge period

Consent:

Patient will be provided with a patient information sheet and have a minimum of one hour to consider trial participation. A longer period for consideration of trial participation can be provided if required by the patient, however baseline assessments must be made within 16 hours of hospital admission.

Risk and benefit:

Sticker placement for the EMG electrodes may require participants to shave their chest. The adhesive stickers and the skin preparation gel may cause minor skin irritation. Participants are required to perform sniff manoeuvres as part of NRD measurement which may feel uncomfortable. Participants will be advised to breath normally should they feel light headed or breathless.

There will be no direct benefit to individual participants. However the study aims to develop a technique that can be used to predict and prevent hospital readmission following admission with exacerbation of COPD, which will have benefits for the wider community of patients and the NHS.

Confidentiality:

Participants' name, date of birth and other identifiable information will be collected during the study phase. All stored data will be in line with the Caldicott principals, data protection and REC guidelines.

Conflicts of interest:

There are no perceived conflicts of interest. Participants' supervising consultants will remain responsible for clinical care and will not be involved in the collection or interpretation of the research data, which will be performed by a dedicated research team.

Tissue and biological samples:

No tissue or biological samples will be obtained for the study protocol outside of routine care.

Protocol amendments:

In September 2018, the following amendments were made to the protocol which were approved by the London-Westminster Research Ethics Committee:

* Addition of the Modified Borg Score to daily assessments to measure subjective breathlessness intensity
* Inclusion criterion six was amended so that participants must live in the catchment area served by the Integrated Respiratory Team (not the "Lane Fox Respiratory Unit") at Guy's and St Thomas' NHS Foundation Trust for clinical, safety and practical purposes.
* Collection of hospital admission, healthcare utilisation and mortality data following study participation from electronic medical records

ELIGIBILITY:
Inclusion Criteria:

* Age 40-80 years
* Patients hospitalized with a primary diagnosis of an acute exacerbation of COPD
* Body mass index (BMI) ≤ 35 kg/m2
* Cognitively and linguistically able to follow instructions given in English and provide informed consent
* To be discharged to home following the hospitalization
* Patient lives in the catchment area served by the Integrated Respiratory Team at Guy's and St Thomas' NHS Foundation Trust in a home environment deemed safe by the investigators to perform home assessments

Exclusion Criteria:

* Previous home PAP (CPAP or NIV) therapy use within the past year, or post-discharge
* Allergies to latex, metals or local anaesthetic agents
* Wound or inflamed skin at parasternal location (2nd intercostal space)
* History of skin allergies or sensitivity to cosmetics and lotions
* Psychological and social factors that would impair compliance with study protocol and schedule
* Any major non-COPD chronic disease or condition, such as severe heart failure (LVEF<30%), malignancy (active treatment and palliation), end stage renal failure/dialysis, significant neuromuscular disease (e.g. NMD, MD) determined by review of medical history and / or patient reported medical history that may contribute significantly to risk of readmission, as determined by PI
* Length of stay ≤ 24 hours
* Planned travel away from home within the 30 day post discharge period

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to hospital with a primary diagnosis of an acute exacerbation of COPD.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
Change in NRD from baseline to day prior to an acute exacerbation of COPD. | 30 days
  Change in EMGpara%max (derived from RMS EMGpara and maximal sniff manoevres) from subjects' baseline NRD to the day before a clinical re-exacerbation of COPD following index hospitalisation with AECOPD.

SECONDARY OUTCOMES:
Change in NRD from peak exacerbation (hospital) to recovery baseline (home) | 30 days
  Change in NRD (measured as EMGpara%max) from its peak during hospital admission to baseline which will occur during the recovery period at home.
Correlation of time to recovery as measured by NRD and EXACT-PRO | 30 days
  Time to recover NRD from hospital peak to home baseline will be correlated with EXACT-PRO score. The EXACT-PRO score is designed to standardize the method for evaluating the frequency, severity and duration of both reported and unreported AECOPD in studies. The EXACT-PRO total score is computed across the 14 items and has a theoretical range of 0 to 100, with higher values indicating a more severe condition. Specifically, the changes in the total score may be used to define recovery from the primary exacerbation event.
Correlation of NRD to EXACT-PRO from hospital discharge to recovery | 30 days
  NRD measurements will be compared to EXACT-PRO questionnaire scores to examine for a correlation between patient-reported symptoms and NRD.
Correlation of NRD to physical activity from hospital discharge to recovery | 30 days
  NRD measurements will be compared to physical activity to examine for a correlation between physical activity and sleep-wake cycle and NRD. This correlation will be examined to evaluate physical activity as an additional advanced physiological biomarker to identify further re-exacerbations of COPD and predict readmission. It will be measured using physical activity monitors which are wrist-worn devices. Using an accelerometer, the physical activity monitor will collect data on total sleep time, time spent awake after sleep onset, sleep onset latency, sleep efficiency, average activity (counts/minute), maximum activity (counts/minute), mobile time, average mobile bout, immobile time and total wake and sleep times.
Physician-assessed exacerbation within 30-day post-discharge | 30 days
  Defined as "worsening respiratory symptoms (cough, wheeze, increased sputum production, increased volume of sputum and/or increased breathlessness) with physician assessment and COPD treatment escalated (increased beta-agonist use as inhaled or nebulized therapy and/or oral corticosteroids and/or oral antibiotics) by physician WITHOUT admission to hospital". This data will be obtained from medical records and participants' symptom diaries.
Self-treated exacerbation within 30-day post-discharge | 30 days
  Defined as "worsening respiratory symptoms (cough, wheeze, increased sputum production, increased volume of sputum and/or increased breathlessness) WITHOUT physician assessment but patient self-initiated AECOPD treatment (use of rescue pack of oral corticosteroids and/or oral antibiotics, depending on standard of care at clinical site)". This data will be obtained from participants' symptom diaries.
All cause hospital readmission within 30-day post-discharge | 30 days
  This data will be collected from electronic medical records.
Mortality within 30-day post-discharge | 30 days
  This data will be collected from electronic medical records and by contacting participants' primary care physicians if necessary.
Recovery as defined by the EXACT-PRO within 30-day post-discharge | 30 days
  Use of the EXACT-PRO score to identify time to recovery within the 30-day post-discharge period.
Medication change within 30-day post-discharge | 30 days
  Use of participants' symptom diary to identify COPD medication changes within 30-day post-discharge.
Unplanned healthcare contacts | 30 days
  Use of participants' symptom diaries and medical records to evaluate healthcare utilization in the 30-day post-discharge period.
Attendance of emergency department (without admission) | 30 days
  Use of participants' symptom diaries and medical records to evaluate healthcare utilization in the 30-day post-discharge period.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Hart, MBBSPhDFFICM, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guys and St Thomas NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2017-09-04): https://cdn.clinicaltrials.gov/large-docs/05/NCT03443505/Prot_000.pdf
  • Informed Consent Form (2017-09-04): https://cdn.clinicaltrials.gov/large-docs/05/NCT03443505/ICF_001.pdf